CLINICAL TRIAL: NCT03126305
Title: Facilitating Fidelity and Dissemination of Evidence Based Treatment for Childhood OCD Via an Interactive Crowd-sourced Patient-provider Tool
Brief Title: Initial Development and Dissemination of OC-Go
Acronym: OC-GoPhaseI
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Virtually Better, Inc. (Industry)
Responsible Party: Principal Investigator, John Piacentini, Professor of Psychiatry and Biobehavioral Sciences, University of California, Los Angeles
Other Study IDs: R42MH111277-01A1 (NIH)
Record Dates: First submitted 2017-04-19; First posted 2017-04-24 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: exposure; response prevention; web-based application
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OC-Go: Approximately 10-20 9-17 year-olds receiving exposure based cognitive behavior therapy for OCD through the UCLA Division of Child and Adolescent Psychiatry OCD treatment programs
  Interventions: Other: OC-Go

INTERVENTIONS:
Other: OC-Go — OC-Go, a HIPAA-compliant web-based clinician portal and patient-side mobile application that allows clinicians to create and push tailored treatment assignments to patients on their mobile devices

SUMMARY:
The clinical component of Phase I application development examines the clinical utility, feasibility, and functionality of the OC-Go application via an 8-month pilot trial consisting of 50 standard CBT sessions augmented with OC-Go in OCD-diagnosed children who are receiving treatment through the pediatric OCD treatment programs in the UCLA Division of Child and Adolescent Psychiatry

DETAILED DESCRIPTION:
This project seeks to refine and assess OC-Go, a HIPAA-compliant web-based clinician portal and patient-side mobile application designed to increase patient adherence to evidence-based treatment (EBT) for Obsessive Compulsive Disorder (OCD), a common and impairing condition, and provider ability to effectively implement EBTs. OC-Go allows clinicians to create and push tailored assignments to patients on their mobile devices with an optimized user interface that includes patient accountability and support features. Accordingly, patients can be guided to do assignments by themselves between sessions with increased fidelity over the course of treatment. Once therapy assignments are created and shared to a crowd-sourced and curated public library, any clinician can assign any task to any patient for homework or in-session use with one touch. Use of OC-Go is expected to increase patient engagement, compliance, treatment efficiency, dissemination of EBTs, and therapist confidence and expertise.

ELIGIBILITY:
Inclusion Criteria:

* Children receiving exposure based CBT through the UCLA Child OCD, Anxiety and Tic Disorders Clinic or Pediatric OCD Intensive Outpatient Program and their parents

Exclusion Criteria:

* None

Ages: 9 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children receiving exposure based CBT through the UCLA Child OCD, Anxiety and Tic Disorders Clinic or Pediatric OCD Intensive Outpatient Program and their parents
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
System Usability Scale (SUS) | 6 weeks
  10-item self-report measure assessing the usability of the OC-Go application
Usability Evaluation for e-Learning Applications (UELA), | 6 weeks
  54-item self-report measure assessing the usability of the OC-Go application

CONTACTS AND LOCATIONS:
Overall Officials: John Piacentini, Ph.D., Principal Investigator — University of California, Los Angeles; Peter Tuerk, Ph.D., Principal Investigator — Virtually Better, Inc.
Locations (1):
- Univ. of California / Los Angeles / Semel Inst., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No